CLINICAL TRIAL: NCT03928431
Title: Restoration of Microbiota in Neonates - a Randomized Controlled Trial
Brief Title: Restoration of Microbiota in Neonates
Acronym: RoMaNs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other); Linkoeping University (Other Government); Umeå University (Other); Örebro University, Sweden (Other); Jonkoping University (Other)
Responsible Party: Principal Investigator, Lars Engstrand, professor, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/1298-31/1
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis; Atopic Asthma; Immunologic Activity Alteration
Keywords: microbiota; cesarean section; vaginal delivery; allergy; immunological programming
MeSH Terms: conditions — Dermatitis, Atopic; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: In this RCT, 330 infants of healthy mothers (age 18 to 40 years) with uncomplicated pregnancies will be included and the infants followed primarily for two years. The number has been increased to cover for potential drop-outs.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Mothers who give birth by CS will be randomized to expose their neonate to samples of their vaginal and fecal microbiome after birth or to placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- vaginally delivered (No Intervention): A non-randomized reference group of vaginally delivered infants.
- CS intervention (Active Comparator): A piece of gauze soaked with saline (0.9%) will be placed in the birth canal 2 hours before the CS by the study midwife, using sterile glows. Before the CS procedure begins, the gauze will be removed from the vagina and then immediately "contaminated" by a swab carrying maternal fecal microbiota. The swab is contaminated by introducing it 3 cm into the anal canal and by rotating it for 10-20 s.
  Immediately after birth, the study midwife will swab the neonate with the gauze in multiple body sites by a standardized manner and then swab maternal breasts and chest skin. The neonate will then be placed on the maternal chest to initiate breast-feeding.
  Interventions: Other: Maternal microbiota
- CS placebo (Placebo Comparator): See above - the gauze will be exchanged to a clean gauze (soaked with saline). Immediately after birth, the study midwife will swab the neonate with the gauze in multiple body sites by a standardized manner and then swab maternal breasts and chest skin. The neonate will then be placed on the maternal chest to initiate breast-feeding.
  Interventions: Other: Maternal microbiota

INTERVENTIONS:
Other: Maternal microbiota — See arm descriptions
  Arms: CS intervention; CS placebo

SUMMARY:
The aim of the study is to examine the effect of exposure of cesarean section (CS) delivered neonates to a natural condition of birth, i.e. to the microbiota of the birth canal, on the acquisition of microbial genes during development of the microbiome at multiple body sites, immune system maturation and allergy risk in childhood

DETAILED DESCRIPTION:
The primary outcome is to examine if exposure to the maternal vaginal and fecal microbiota directly after birth will halfen the cumulative incidence of Immunoglubulin E (IgE)-associated allergic disease at 2 years of age in CS delivered infants, compared with non-treated CS-delivered infants.

The secondary outcomes are to compare the community structure of microbes from mothers and their infants and immunological programming of infants delivered via scheduled CS, with or without exposure to the maternal vaginal and fecal microbiota, from birth until two years of age. The primary and secondary outcomes will also be compared with a reference group of vaginally delivered infants. Sex differences in the incidence and prevalence of allergic diseases have been described. The anticipated benefit of the intervention can be implemented in clinical practice regardless of sex, so that improved conditions for good health are created.

ELIGIBILITY:
Inclusion Criteria:

* Infants of healthy mothers with uncomplicated pregnancies at term, mothers of any ethnic or social background that can speak, read, and understand Swedish to the extent that they can consent in Swedish. An additional inclusion criterion for mothers in the CS groups is vaginal pH ≤ 4 at the time of birth.

Exclusion Criteria:

* Infants of mothers with pre-eclampsia or complicated pregnancies, mothers <18 years or >40 years of age, genital herpes simplex, genital warts, HIV, Hepatitis B or complications during delivery, infants delivered prior to 37 weeks of gestation. Additional exclusion criteria for mothers in the CS group: Mothers positive to Group B Streptococcus, Group A Streptococcus, bacterial vaginosis, vaginal pH > 4 at the time of birth. Mothers with fecal samples positive for Salmonella, Shigella, Campylobacter or Yersinia.

Ages: 5 Minutes to 15 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
IgE-associated allergic disease | Two years
  Incidence of Immunoglubulin E (IgE)-associated allergic disease at 2 years of age in CS delivered infants, compared with non-treated CS-delivered infants and vaginally delivered controls.
  Skin-puncture tests will be performed at infant age 6 months, 12 months and child age 24 months.

SECONDARY OUTCOMES:
Immunological programming | Two years
  Immunological programming will be assessd via blood cell count from blood tests at 6,12 nad 24 months in infants delivered via scheduled CS, with or without exposure to the maternal vaginal and fecal microbiota in comparison to infants born vaginally.
Development of the microbiota | Two years
  To compare microbial composition between groups, using shotgun metagenomics.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Nylén, PhD, Study Chair — Dept Microbiology, Tumour and Cell Biology, Karolinska Institutet, Stockholm
Locations (1):
- Karolinska Institutet, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Samples will be stored at Karolinska Biobank and metadata will be linked to these samples with access for all researchers in the study. No data will be available for researchers outside the consortium.